CLINICAL TRIAL: NCT07081529
Title: Clinical Evaluation of Direct and Indirect Restorations in Class I Cavities: A 10-Year Follow-up Study
Brief Title: Clinical Evaluation of Class I Direct and Indirect Restorations Over 10 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Neslihan Tekçe, Professor Dr., Kocaeli University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/157
Record Dates: First submitted 2025-07-10; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Clinical Trial; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Direct and Indirect Restorations (Experimental): Participants in this arm received two different types of restorations in Class I cavities of molar teeth: one direct restoration using a microhybrid universal composite, and one indirect restoration using a reinforced microfill composite system. Each patient received one of each restoration type on different molar teeth. Clinical evaluations were conducted at baseline, 1 year, 2 years, and 10 years using modified USPHS criteria.
  Interventions: Device: Direct Restoration with Microhybrid Composite; Device: Indirect Restoration with Reinforced Microfill Composite

INTERVENTIONS:
Device: Direct Restoration with Microhybrid Composite — Direct Class I restorations were placed in molar teeth using a microhybrid universal composite (Aelite All-Purpose Body, Bisco) and an adhesive system according to the manufacturer's instructions.
Device: Indirect Restoration with Reinforced Microfill Composite — Indirect Class I restorations were fabricated using a reinforced microfill composite system (Tescera Indirect Composite System Body, Bisco) in the laboratory and cemented into molar teeth using resin cement.

SUMMARY:
This clinical study aims to evaluate and compare the long-term clinical performance of direct and indirect restorations in Class I cavities of molar teeth over a 10-year period. A total of 54 restorations (27 direct and 27 indirect) were placed in 27 patients, with each patient receiving one direct and one indirect restoration. The restorations were evaluated at baseline, and at 1-, 2-, and 10-year follow-ups using modified USPHS criteria.

DETAILED DESCRIPTION:
This prospective clinical study was designed to evaluate and compare the long-term clinical performance of direct and indirect composite restorations in Class I cavities of permanent molar teeth over a 10-year period.

A total of 27 patients were enrolled in the study. Each participant received one direct and one indirect restoration, resulting in a total of 54 restorations (27 direct and 27 indirect).

Direct restorations were performed intraorally using a microhybrid composite and adhesive system in accordance with the manufacturer's instructions. Indirect restorations were fabricated in the laboratory using a reinforced microfill composite system and cemented using resin cement.

All restorations were clinically evaluated at baseline, and at 1-, 2-, and 10-year follow-up appointments. The modified United States Public Health Service (USPHS) criteria were used for evaluation. The assessed parameters included surface texture, anatomic form, color match, marginal adaptation, cavosurface marginal discoloration, and the presence of caries.

The aim of this study is to provide evidence-based clinical data regarding the durability and performance of direct and indirect composite restorations in posterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with two Class I cavities
* Good oral hygiene maintenance
* Absence of pulp or periodontal disease
* Requirement for restoration of permanent molars due to occlusal caries

Exclusion Criteria:

* Presence of parafunctional habits (e.g., bruxism or clenching)
* Poor oral hygiene
* Lack of interest in or refusal to comply with oral hygiene instructions
* Pulp exposure during caries removal
* Percussion sensitivity indicating possible pulpal or periapical pathology
* Spontaneous discomfort associated with periodontal disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
10-Year Clinical Success Rate of Direct and Indirect Restorations | 10 years
  The primary outcome is the clinical success rate of direct and indirect Class I restorations in molar teeth after 10 years. Success and failure were assessed using modified United States Public Health Service (USPHS) criteria. A restoration was considered a failure if it required replacement due to secondary caries or other clinical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Tekçe, Principal Investigator — Kocaeli University, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tekce N, Demirci M, Tuncer S, Oghan Turkoglu M, Turgut V, Balci SN, Yersel G. Clinical evaluation of direct and indirect restorations in class I cavities: a 10-year follow-up study. BMC Oral Health. 2025 Sep 25;25(1):1430. doi: 10.1186/s12903-025-06775-9. PMID 40999454